CLINICAL TRIAL: NCT07021248
Title: A Randomized Controlled Trial Evaluating the Impact of Procedure-Specific Bariatric Supplements on Micronutrient Status and Vitamin B6 Hypervitaminosis Following Metabolic and Bariatric Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: General Committee of Teaching Hospitals and Institutes, Egypt (Other Government)
Responsible Party: Principal Investigator, Mohamed Hany Ashour, Professor of General surgery, General Committee of Teaching Hospitals and Institutes, Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RCT Micronutrient Status
Record Dates: First submitted 2025-05-26; First posted 2025-06-13 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Micronutrient Status
Keywords: Procedure-Specific Bariatric Supplements; Micronutrient Status; Vitamin B6 Hypervitaminosis; Metabolic and Bariatric Surgery

STUDY DESIGN:
Intervention Model Description: Participants will receive a specialized Elan bariatric supplement matched to the type of MBS they undergo. Each formulation, Elan Believe for SG, Elan Compass for RYGB, and Elan Supreme for OAGB, addresses the distinct micronutrient absorption profiles and physiological alterations associated with each surgical procedure. Importantly, all three formulations contain a standardized dose of vitamin B6 of 400 micrograms, facilitating valid comparisons of postoperative B6 levels across procedures.
  Supplementation will commence after one month postoperatively and continue for 12 months. Participants will be instructed to take one tablet daily with food. In addition to the assigned Elan supplement, all participants will receive standard calcium and cholecalciferol supplementation per institutional protocols.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Elan Believe (Active Comparator): Sleeve gastrectomy specific bariatric supplement
  Interventions: Dietary Supplement: Elan Believe
- Elan Compass (Active Comparator): Roux en Y gastric bypass specific bariatric supplement
  Interventions: Dietary Supplement: Elan Compass
- Elan Supreme (Active Comparator): One anastomosis gastric bypass specific bariatric supplement
  Interventions: Dietary Supplement: Elan Supreme

INTERVENTIONS:
Dietary Supplement: Elan Believe — Participants will receive a specialized Elan bariatric supplement matched to the type of MBS they undergo. Elan Believe for SG addresses the distinct micronutrient absorption profiles and physiological alterations associated with this surgical procedure. Importantly, all formulations contain a standardized dose of vitamin B6 of 400 micrograms, facilitating valid comparisons of postoperative B6 levels across procedures.
  Arms: Elan Believe
Dietary Supplement: Elan Compass — Participants will receive a specialized Elan bariatric supplement matched to the type of MBS they undergo. Elan Compass for RYGB addresses the distinct micronutrient absorption profiles and physiological alterations associated with this surgical procedure. Importantly, all formulations contain a standardized dose of vitamin B6 of 400 micrograms, facilitating valid comparisons of postoperative B6 levels across procedures.
  Arms: Elan Compass
Dietary Supplement: Elan Supreme — Participants will receive a specialized Elan bariatric supplement matched to the type of MBS they undergo. Elan Supreme for OAGB addresses the distinct micronutrient absorption profiles and physiological alterations associated with this surgical procedure. Importantly, all formulations contain a standardized dose of vitamin B6 of 400 micrograms, facilitating valid comparisons of postoperative B6 levels across procedures.
  Arms: Elan Supreme

SUMMARY:
Obesity is a complex, multifactorial chronic disease with an escalating global incidence, impacting over 650 million adults worldwide. It is closely linked to a variety of metabolic, cardiovascular, and musculoskeletal diseases, and is a leading contributor to preventable morbidity and mortality. Metabolic and Bariatric Surgery (MBS) stands out as the most effective long-term intervention for obesity, facilitating significant and sustained weight loss while also promoting remission of associated diseases.

However, the anatomical and physiological alterations induced by MBS, including gastric restriction, bypass of absorptive surfaces, altered gastrointestinal transit, and reduced gastric acid production, significantly disrupt nutrient absorption and metabolism, placing patients at lifelong risk of micronutrient deficiencies or, conversely, hypervitaminosis resulting from excessive supplementation. Among these, Vitamin B6 imbalance has emerged as a significant yet under-recognized issue in post-MBS patients.

Among the nutrients affected, vitamin B6 (pyridoxine) presents a unique challenge. Vitamin B6 functions as a coenzyme in amino acid metabolism, neurotransmitter synthesis, and immune regulation. Deficiencies in Vitamin B6 are well-documented and can manifest as glossitis, irritability, and peripheral neuropathy. Notably, B6-related neuropathy may clinically resemble Guillain-Barré syndrome in post-MBS patients. This anxiety surrounding deficiency symptoms often leads to the overconsumption of Vitamin B6, resulting in hypervitaminosis, which can also present with neurological manifestations such as sensory neuropathy and ataxia.

The risk of hypervitaminosis is further exacerbated by the widespread use of high-dose multivitamin formulations post-surgery, many of which contain vitamin B6 at levels far exceeding the Recommended Dietary Allowance (RDA). For males, the RDA is 1.3 mg daily for those aged 19-50 years, increasing to 1.7 mg for those over 50. For females, the RDA is 1.3 mg for those aged 19-50 and 1.5 mg for those over 50. Yet some commercially available bariatric supplements exceed this level several-fold. Studies by Dogan et al. and Homan et al. emphasize the prevalence of vitamin B6 toxicity in post-MBS populations, largely attributable to inappropriate supplementation practices.

DETAILED DESCRIPTION:
To address this, the Elan series of bariatric-specific supplements (Believe, Compass, and Supreme) was developed with standardized and conservative B6 dosing (400 micrograms per day), approximately 29% of the adult RDA. Each formulation is tailored to the nutritional demands of a specific MBS procedure, while maintaining a uniform B6 dose to facilitate direct comparisons of B6 status across surgical types.

To date, no prospective, randomized study has evaluated the effect of procedure-specific supplementation on the risk of vitamin B6 hypervitaminosis in post-bariatric patients. This trial aims to fill that gap by comparing standardized B6 supplementation outcomes across three common MBS procedures: sleeve gastrectomy (SG), Roux-en-Y gastric bypass (RYGB), and one-anastomosis gastric bypass (OAGB).

In addition to assessing the prevalence of B6 toxicity and deficiency, the study will evaluate broader micronutrient status, anthropometric outcomes, and adherence to supplementation. Findings from this trial are expected to inform the design of safer, procedure-matched supplementation protocols for post-MBS care.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants will be adults:

* Aged 18 to 65 years
* Undergoing primary metabolic and bariatric surgery (MBS), including sleeve gastrectomy (SG), Roux-en-Y gastric bypass (RYGB), or one anastomosis gastric bypass (OAGB).
* Patients must meet established surgical indications as defined by the International Federation for the Surgery of Obesity and Metabolic Disorders (IFSO), specifically: a body mass index (BMI) greater than 30 kg/m² with at least one obesity-related comorbidity (e.g., type 2 diabetes, hypertension, obstructive sleep apnea)
* or a BMI greater than 35 kg/m² irrespective of comorbidities.
* Eligible participants must be capable of providing informed consent, willing to adhere to the prescribed supplement regimen, and able to complete scheduled postoperative follow-up visits for 12 months.

Exclusion Criteria:

Exclusion criteria include:

* Revision or secondary MBS procedures
* Known hypersensitivity to vitamin B6 or any component of the supplement formulations
* Pregnancy or planned pregnancy during the study period
* Any pre-existing medical condition known to interfere with vitamin B6 metabolism. This includes, but is not limited to, severe hepatic or renal dysfunction, peripheral neuropathy, and the use of medications such as isoniazid, phenytoin, or levodopa. Additional exclusions include chronic gastrointestinal conditions affecting absorption (e.g., inflammatory bowel disease, celiac disease), porphyria, or any other clinical scenario that, in the judgment of the investigators, may compromise compliance or the reliability of follow-up.
* Patients who are already receiving high-dose vitamin B6 supplementation or have abnormal preoperative B6 levels will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The prevalence of vitamin B6 hypervitaminosis | Measured at 6 and 12 months postoperatively.
  Defined as a serum pyridoxal 5'-phosphate (PLP) concentration greater than 100 nmol/L, measured at 6 and 12 months postoperatively.

SECONDARY OUTCOMES:
Prevalence of vitamin B6 deficiency | Measured at 6 and 12 months postoperatively.
  Defined as a serum PLP concentration less than 25 nmol/L.
Serum concentrations of other key micronutrients | Measured at 6 and 12 months postoperatively.
  Including vitamin B12 (reference range: 150-640 pmol/L), folate, ferritin, zinc, calcium, and parathyroid hormone (PTH)
Incidence of other micronutrient deficiencies | measured at 6 and 12 months postoperatively.
  Including vitamin B12, iron, calcium, folate.
Relationship between supplement adherence and clinical outcomes | measured at 6 and 12 months postoperatively.
  Adherence will be evaluated using: monthly pill counts Associations between adherence levels and biochemical or anthropometric outcomes will be explored using correlation and regression models.
Trends in micronutrient status (hemoglobin, ferritin, vitamin B12, folate, vitamin D, calcium, magnesium, parathyroid hormone, and zinc) | measured at 6 and 12 months postoperatively.
  across the different surgical cohorts (SG, RYGB, and OAGB).
Changes in anthropometric parameters | measured at 6 and 12 months postoperatively.
  including weight (In Kilograms), body mass index (BMI) (weight in kilograms, height in meters) (weight and height will be combined to report BMI in kg/m^2), percentage of excess weight loss (%EWL), and percentage of total weight loss (%TWL)
Relationship between supplement adherence and clinical outcomes | Administered at 6 and 12 months
  Adherence will be evaluated using: the validated 5-item Medication Adherence Report Scale (MARS-5) Questionnaire, administered at 6 and 12 months, a validated instrument that identifies prevalent non-adherence patterns.
  Associations between adherence levels and biochemical or anthropometric outcomes will be explored using correlation and regression models.

CONTACTS AND LOCATIONS:
Locations (1):
- The surgical department of Medical Research Institute Hospital, Alexandria University, Alexandria, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The analysis will be performed on a blinded dataset after completing the medical/scientific review. All protocol violations will be identified and resolved, and the dataset will be declared complete. All data will be collected in a data management system (Castor EDC, Amsterdam, The Netherlands; https://www.castoredc.com), handled according to Good Clinical Practice guidelines, Data Protection Directive certificate, and complied with Title 21 CFR Part 11. Furthermore, the data centers where all the research data will be stored are certified according to ISO27001, ISO9001, and Dutch NEN7510.
  Can be asked by the contact person
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Whole study period
Access Criteria: Ask contact person